CLINICAL TRIAL: NCT01999777
Title: A Randomized, Double-Blind, Placebo Controlled Trial Examining the Safety and Efficacy of Midazolam Intranasal Spray (USL261) for the Treatment of Intermittent Bouts of Increased Seizure Activity in the Epilepsy Monitoring Unit (EMU)
Brief Title: Study to Evaluate the Safety and Efficacy of USL261 in Patients With Increased Bouts of Seizure Activity in the EMU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USL261-301
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; seizure clusters; acute repetitive seizures; rescue treatment
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- USL261 (Experimental): 5 mg intranasal midazolam
  Interventions: Drug: USL261
- Placebo (Placebo Comparator): intranasal placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: USL261
  Arms: USL261
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy, safety, and tolerability of USL261 compared with that of intranasal (IN) placebo for the treatment of intermittent bouts of increased seizure activity.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been admitted to the institution's EMU for seizure characterization or pre-surgical evaluation, or such admission is planned within 28 days
* Subject body weight is ≥ 40 kg to ≤ 125 kg (inclusive)
* Subject has an established diagnosis of partial or generalized epilepsy

Exclusion Criteria:

* Subject has history of status epilepticus in the 6 months prior to Screening
* Subject has a progressive neurological disorder such as brain tumor, demyelinating disease, or degenerative central nervous system (CNS) disease that is likely to progress in the next 12 months
* Subject has respiratory failure (or is at risk for respiratory failure) or other severe cardiorespiratory disease with New York Heart Association Class III or IV functional status, or requires supplemental oxygen
* Subject has acute narrow-angle glaucoma
* Subject is receiving chronic benzodiazepine treatment (defined as an average of ≥ 4 administrations per week) and cannot safely withdraw from such treatment within the washout period prior to treatment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (37):
  - Phoenix, Arizona
  - Tucson, Arizona
  - La Jolla, California
  - Orange, California
  - San Francisco, California
  - Denver, Colorado
  - Englewood, Colorado
  - New Haven, Connecticut
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Winfield, Illinois
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Jackson, Mississippi
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Edison, New Jersey
  - Brooklyn, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Madison, Wisconsin
- Melbourne, Victoria, Australia
- Linz, Austria
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Czechia (2):
  - Brno
  - Prague
- Germany (3):
  - Bonn
  - Kork
  - Tübingen
- Vilnius, Lithuania
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia

REFERENCES:
- [Derived] Spencer DC, Sinha SR, Choi EJ, Cleveland JM, King A, Meng TC, Pullman WE, Sequeira DJ, Van Ess PJ, Wheless JW. Safety and efficacy of midazolam nasal spray for the treatment of intermittent bouts of increased seizure activity in the epilepsy monitoring unit: A double-blind, randomized, placebo-controlled trial. Epilepsia. 2020 Nov;61(11):2415-2425. doi: 10.1111/epi.16704. Epub 2020 Nov 2. PMID 33140403

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 188 eligible subjects entered Pretreatment Observation during which they were monitored in EMU for seizure events. Only subjects who met entry criteria and presented with seizure events meeting the treatment decision criteria were eligible to enter the Treatment Phase. Participant flow represents subjects who took at least 1 dose of study drug.
Groups:
- USL261: 5 mg intranasal midazolam
  USL261
- Placebo: intranasal placebo
  Placebo
Period: Overall Study
Arm/Group | USL261 | Placebo
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refers to the Safety Analysis Set which included all subjects who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | USL261 | Placebo | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (12.94) | 35.9 (13.56) | 34.3 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 26 | 27 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 0 | 1
  United States | 22 | 22 | 44
  Czechia | 2 | 2 | 4
  Lithuania | 3 | 2 | 5
  Germany | 0 | 1 | 1
  Spain | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were Seizure-free
Description: A participant was considered "seizure-free" if he or she completed the 6-hour Treatment Phase without seizures recorded, premature discontinuation of study drug, rescue intervention for acute central respiratory depression adverse event (AE), and alterations to background anti-epileptic drug (AED) therapy. Otherwise, the participant was included in the analysis for seizure-free events with the outcome of "seizure."
Time Frame: 6 hours
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | USL261 | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 17 | 12
Statistical Analysis 1: Comparison: USL261 vs Placebo; Assumptions included that the proportion of seizures occurring within 6 hours after placebo administration was ~65% and a relative reduction of 50% would result in a reduction of ≥ 32.5 percentage points. Based on a 2-sided 95% confidence interval (CI) for the differences in proportions, a sample size of 62 analyzable subjects was chosen to detect a 0.35 difference between group. Sample size estimations were based on nQuery Version 7.0 using the table for CIs for differences in 2 proportions; Test type: Superiority; p = 0.1972, Wald asymptotic; P-value based on a standard Wald asymptotic test for equality without a continuity correction

2. Secondary Outcome: Time to First Seizure Following Treatment (TFSFT)
Description: Time to first seizure following treatment was defined as time from treatment with study drug to the onset of the next seizure, rescue intervention (for acute central respiratory depression AE) to maintain subject safety, alterations to background AED therapy, early termination, or 6 hours, whichever came first.
Time Frame: 6 hours
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | USL261 | Placebo
Number analyzed (Participants) | 31 | 31
hours | NA [4.0 to NA] — Unable to estimate median as > 50% were seizure-free throughout the 6-hour treatment phase. No upper CI boundary as observations stopped at 6 hours. | 3.9 [1.8 to NA] — No upper CI boundary as observations stopped at 6 hours.
Statistical Analysis 1: Comparison: USL261 vs Placebo; Test type: Superiority; p = 0.1388, Log Rank

ADVERSE EVENTS:
Time Frame: From informed consent until up to 48 hours of completion of the Treatment Phase
Description: Adverse events were collected from time of informed consent until subject completion or early termination. Exit assessments were to be conducted within 48 hours of completion of the Treatment Phase (6 hours) and prior to discharge for the EMU.
Arm/Group | USL261 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 16/31 | 17/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | USL261 (N=31) | Placebo (N=31)
Nausea (Gastrointestinal disorders) | 3 | 1
Product taste abnormal (General disorders) | 2 | 6
Rhinitis (Infections and infestations) | 0 | 2
Tongue injury (Injury, poisoning and procedural complications) | 0 | 2
Headache (Nervous system disorders) | 1 | 5
Somnolence (Nervous system disorders) | 2 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A manuscript or abstract should not be submitted by investigator(s) for publication or presentation until a New Drug Application is approved by the US FDA or permission is granted in writing by the sponsor.